CLINICAL TRIAL: NCT05364645
Title: A Randomized Phase II Study of Carboplatin and Pemetrexed w/ or w/o Selpercatinib in Participants With Non-Squamous RET Fusion-Positive Stage IV Non-Small Cell Lung Cancer and Progression of Disease on Prior RET Directed Therapy (Lung-MAP Sub-Study)
Brief Title: Testing the Use of Targeted Treatment for RET Positive Advanced Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S1900F; NCI-2022-02517 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1900F (Other: SWOG); S1900F (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Carboplatin; Pemetrexed; selpercatinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (carboplatin, pemetrexed, selpercatinib) (Experimental): Patients receive carboplatin IV over 30 minutes and pemetrexed IV over 10 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also selpercatinib PO BID in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Selpercatinib
- Arm B (carboplatin, pemetrexed) (Active Comparator): Patients receive carboplatin IV over 30 minutes and pemetrexed IV over 10 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
Drug: Selpercatinib — Given PO
  Other Names: LOXO-292; RET Kinase Inhibitor LOXO-292; Retevmo; WHO 10967
  Arms: Arm A (carboplatin, pemetrexed, selpercatinib)

SUMMARY:
This phase II Lung-MAP treatment trial tests whether carboplatin and pemetrexed with or without selpercatinib works to shrink tumors in patients with RET fusion-positive non-small cell lung cancer that is stage IV or has not responded to previous RET directed therapy. Chemotherapy drugs, such as carboplatin and pemetrexed, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Selpercatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving selpercatinib in combination with carboplatin and pemetrexed may help lower the chance of the cancer growing and spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare investigator-assessed progression-free survival (IA-PFS) in participants with RET fusion-positive non-small cell lung cancer (NSCLC) with acquired selective RET inhibitor resistance randomized to carboplatin and pemetrexed with or without selpercatinib.

SECONDARY OBJECTIVES:

I. To evaluate if the combination of selpercatinib combined with carboplatin and pemetrexed during the first cycle of treatment has an acceptable toxicity rate.

II. To evaluate the frequency and severity of toxicities within the arms. III. To compare the investigator-assessed objective response rate (ORR) (complete or partial confirmed response) between the arms.

IV. To compare overall survival (OS) between the arms. V. To evaluate duration of investigator-assessed response among responders within each treatment arm.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To collect, process, and bank cell-free deoxyribonucleic acid (cfDNA) at baseline, progression, and end of treatment for future development of a proposal to evaluate comprehensive next-generation sequencing of circulating tumor deoxyribonucleic acid (ctDNA).

II. To establish a tissue/blood repository from participants with refractory non-small cell lung cancer (NSCLC).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive carboplatin intravenously (IV) over 30 minutes and pemetrexed IV over 10 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also selpercatinib orally (PO) twice daily (BID) in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive carboplatin IV over 30 minutes and pemetrexed IV over 10 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients who had disease progression are followed up every 6 months for 2 years and then at 3 years. Patients who did not have disease progression are followed up every 12 weeks until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have stage IV or recurrent disease
* Participants must have been assigned to S1900F based on biomarker analysis of tissue and/or blood and determined to have RET fusion-positive NSCLC as defined here:

  * Participants must have RET fusion-positive NSCLC as determined by the Foundation Medicine (FMI) tissue-assay or other tumor-based assays such as next generation sequencing (NGS), polymerase chain reaction (PCR), or fluorescent in situ hybridization (FISH), or by cfDNA blood assay as outlined in the LUNGMAP Screening Protocol. Participants previously tested for and determined to have RET-fusion-positive NSCLC outside of LUNGMAP, must also submit tissue for central FMI testing on the LUNGMAP Screening Protocol. Participants with RET fusions detected by IHC alone are not eligible. The testing must be done within a laboratory with Clinical Laboratory Improvement Act (CLIA), International Organization for Standardization (ISO)/International Electrotechnical Commission (IEC), College of American Pathologists (CAP), or similar certification. Presence of RET fusions detected on tests performed outside of LUNGMAP must have been confirmed by the study biomarker review panel
* Participants must be negative for all additional validated oncogenic drivers that could cause resistance to selpercatinib treatment. This includes EGFR sensitizing mutations, EGFR T790M mutations, ALK gene fusions, ROS1 gene fusion, KRAS activating mutations, BRAF V600E mutation and MET exon 14 skipping mutations or high-level amplification and expression

  * NOTE: EGFR, ALK, ROS, KRAS, and BRAF testing is performed as part of the LUNGMAP screening/pre-screening FoundationOne test. If prior data is not available, results from the FMI testing must be obtained prior to sub-study randomization.
* Participants must have measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI). The CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality. Measurable disease must be assessed within 28 days prior to sub-study randomization. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non-measurable disease must be assessed within 42 days prior to sub-study randomization. All disease must be assessed and documented on the Baseline Tumor Assessment Form. Participants whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to randomization
* Participants must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to sub-study randomization
* Participants must have received and developed disease progression during or after an anti-RET inhibitors treatment. The anti-RET inhibitor therapy must be the most recent therapy
* Participants must have progressed (in the opinion of the treating physician) following the most recent line of therapy
* Participants must have recovered (=< grade 1) from any side effects of prior therapy. Participants must not have received any radiation therapy within 14 days prior to sub-study randomization
* For participants with stage IV or recurrent disease, the participant must not have received a platinum-based chemotherapy regimen. For participants whose prior systemic therapy was for stage I-III disease only (i.e., participant has not received any treatment for stage IV or recurrent disease), disease progression on platinum-based chemotherapy must not have occurred within one year (365 days) from the last date that the participant received that therapy. Prior anti-PD-1/PD-L1 therapy, alone or in combination (e.g., nivolumab, pembrolizumab, or durvalumab) is allowed
* Participants must have an electrocardiogram (ECG) performed within 28 days prior to sub-study randomization. It is suggested that a local cardiologist review the corrected QT by Fridericia's correction formula (QTcF) intervals
* Absolute neutrophil count (ANC) >= 1.5 x 10^3/uL obtained within 28 days prior to sub-study randomization
* Platelet count >= 100 x 10^3/uL obtained within 28 days prior to sub-study randomization
* Hemoglobin >= 9 g/dL obtained within 28 days prior to sub-study randomization
* Serum bilirubin =< institutional upper limit of normal (IULN) and either alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 2 x IULN within 28 days prior to sub-study randomization (if both ALT and AST are done, both must be < 2 x IULN). For participants with liver metastases, bilirubin and either ALT or AST must be =< 5 x IULN (if both ALT and AST are done, both must be =< 5 x IULN)
* Participants must have a serum creatinine =< the IULN OR measured or calculated creatinine clearance >= 50 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to sub-study randomization
* Participants must have Zubrod performance status 0-1 documented within 28 days prior to sub-study randomization
* Participants must provide pre-study history and physical exam within 28 days prior to sub-study randomization
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on suppressive therapy within 28 days prior to sub-study randomization
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment must have an undetectable HCV viral load within 28 days prior to sub-study randomization
* Participants with known human immunodeficiency virus (HIV) infection are eligible, provided they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 6 months prior to sub-study randomization
* Participants must be able to swallow capsules
* Participants must agree to have blood specimens submitted for circulating tumor DNA (ctDNA)
* Participants must also be offered participation in banking and in the correlative studies for collection and future use of specimens
* Participants with impaired decision-making capacity are eligible as long as their neurological or psychological condition does not preclude their safe participation in the study (e.g., tracking pill consumption and reporting adverse events to the investigator)
* Participants must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Participants must not have leptomeningeal disease, spinal cord compression or brain metastases unless: (1) metastases have been locally treated and have remained clinically controlled and asymptomatic for at least 14 days following treatment, and prior to sub-study randomization, AND (2) participant has no residual neurological dysfunction and has been off corticosteroids for at least 24 hours prior to sub-study randomization
* Participants must not have received any prior systemic therapy (systemic chemotherapy, tyrosine kinase inhibitor [TKI], immunotherapy or investigational drug) within 14 days prior to sub-study randomization
* Participants must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment while receiving treatment on this study. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not have had a major surgery within 14 days prior to sub-study randomization. Participants must have fully recovered from the effects of prior surgery in the opinion of the treating investigator
* Participants must not have any grade III/IV cardiac disease as defined by the New York Heart Association Criteria (i.e., participants with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within 6 months, or serious uncontrolled cardiac arrhythmia
* Participants must not be pregnant or nursing. Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-25 (Estimated); Primary Completion 2023-06-27 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed progression-free survival (PFS) | From date of sub-study randomization to date of first documentation of progression assessed by local review or symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Will be compared between the arms using a 1-sided log-rank test at the 0.10 level upon the observation of 55 PFS events or at a maximum follow-up duration (from closure of accrual of 15 months). Will be estimated using the method of Kaplan-Meier. Confidence intervals about median event times will be estimated using the Brookmeyer-Crowley method. For point estimates at landmark times, the associated 95% confidence interval (CI) will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. Hazard ratios for these outcomes will be estimated using a Cox Proportional Hazards regression.

SECONDARY OUTCOMES:
Incidence of grade 3 or higher non hematologic toxicity and grade 4 or higher hematologic toxicity | During first cycle (1 cycle = 21 days)
Frequency and severity of adverse events | Up to 3 years
Investigator-assessed objective response rate | Up to 3 years
Overall survival | From date of sub-study randomization to date of death due to any cause, assessed up to 3 years
  Will be estimated using the method of Kaplan-Meier. Confidence intervals about median event times will be estimated using the Brookmeyer-Crowley method. For point estimates at landmark times, the associated 95% CI will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. Hazard ratios for these outcomes will be estimated using a Cox Proportional Hazards regression.
Duration of investigator-assessed response | From date of first documentation of response (complete response [CR] or partial response [PR]) to date of first documentation of progression, or death due to any cause among participants who achieve a response (CR or PR), assessed up to 3 years
  Will be estimated using the method of Kaplan-Meier. Confidence intervals about median event times will be estimated using the Brookmeyer-Crowley method. For point estimates at landmark times, the associated 95% CI will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. Hazard ratios for these outcomes will be estimated using a Cox Proportional Hazards regression.

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Y Elamin, Principal Investigator — SWOG Cancer Research Network
Locations (265):
- United States (265):
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Saint Helena Hospital, St. Helena, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - HaysMed University of Kansas Health System, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - UPMC Western Maryland, Cumberland, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Camp Hill, Camp Hill, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant - Cranberry, Cranberry Township, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Oncology Hematology Associates, Greenville, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - UPMC West Mifflin-Cancer Center Jefferson, West Mifflin, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin